CLINICAL TRIAL: NCT04331314
Title: Sinus Augmentation Using Symbios Versus Algipore as Bone Graft Material - A Randomized Controlled Clinical Pilot Study
Brief Title: Biphasic Calcium Phosphate vs. Hydroxyapatite in Sinus Floor Elevation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27-224 ex 14/15
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Bone Substitutes; Calcium Phosphates; Hydroxyapatite; Rhodophyta; Sinus Floor Augmentation

STUDY DESIGN:
Intervention Model Description: Twenty patients scheduled for lateral-window sinus floor Elevation SFE will be randomized to an HA and a β-TCP/HA Group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SYMBIOS® (Experimental): Sinus augmentation with SYMBIOS® Biphasic Bone Graft Material
  Interventions: Device: Use of Symbios Bone Graft Material
- Algipore® (Active Comparator): Sinus augmentation with Algipore® Bone Substitution Material
  Interventions: Device: Algipore Bone Substitution Material

INTERVENTIONS:
Device: Use of Symbios Bone Graft Material — Patients will receive Symbios Bone Graft Material according to randomization Group.
  Arms: SYMBIOS®
Device: Algipore Bone Substitution Material — Patients will receive Algipore Bone Substitution Material according to randomization Group.
  Arms: Algipore®

SUMMARY:
Twenty patients scheduled for lateral-window sinus floor Elevation (SFE) are randomized into two groups: use of SYMBIOS® Biphasic Bone Graft Material (Group 1) or of Algipore® Bone Substitution Material (Group 2).

Biopsies are taken 3 months after SFE and during implant surgery after 6 months. One ground section per biopsy (n=40) is stained, scanned, and histomorphometrically analyzed for new bone, old bone, soft tissue, graft, bone infiltration of graft, bone-to-graft contact, and penetration depth.

ELIGIBILITY:
Inclusion Criteria:

1. Capability of giving an informed consent
2. Good health as defined by the subject's medical history
3. Patients age 20-75 years
4. Fully edentulous or partially edentulous patients with unilateral or bilateral missing teeth in the maxillary premolar or molar areas with severe alveolar atrophy and a residual alveolar ridge height of maximal 5 mm requiring a two-staged sinus floor elevation and implant placement.

Exclusion Criteria:

1. Patients without detailed baseline medical data
2. Patients with medical history of local inflammations in the posterior maxilla
3. Skeletal immaturity
4. Patients with osteoporosis in their medical history
5. Patients with severe illnesses, malignant diseases, radiotherapy or chemotherapy in their medical history
6. Patients with pathological fractures
7. Patients treated with bisphosphonates
8. Uncontrolled diabetes mellitus
9. Uncontrolled periodontal diseases
10. Smoking
11. Pregnancy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Implant stability | 12 months after sinus augmentation
  measured with Periotest®

SECONDARY OUTCOMES:
Survival rate of the implants | 24 months after sinus augmentation
  Rate of loss of implants
Probing on depth | 24 months after sinus augmentation
  The measurement of probing depth will be performed with a CPITN probe with 0.5mm ball head
Bleeding on probing | 24 months
Crestal bone level after implant | 12 months after implant placement
  measured by means of single tooth x-rays
Complications | 6 months after sinus augmentation
  Frequency of complications
Newly formed bone area in mm² | 3 months after sinus augmentation
  measured through histomorphological analysis
Newly formed bone area in mm² | 6 months after sinus augmentation
  measured through histomorphological analysis
Old bone area in mm² | 3 months after sinus augmentation
  measured through histomorphological analysis
Old bone area in mm² | 6 months after sinus augmentation
  measured through histomorphological analysis
Tissue area in mm² | 3 months after sinus augmentation
  measured through histomorphological analysis
Tissue area in mm² | 6 months after sinus augmentation
  measured through histomorphological analysis
Bone substitute area in mm² | 3 months after sinus augmentation
  measured through histomorphological analysis
Bone substitute area in mm² | 6 months after sinus augmentation
  measured through histomorphological analysis
New bone infiltration area in bone substitute in mm² | 3 months after sinus augmentation
  measured through histomorphological analysis
New bone infiltration area in bone substitute in mm² | 6 months after sinus augmentation
  measured through histomorphological analysis
new bone to bone substitute contact in mm | 6 months after sinus augmentation
  measured through histomorphological analysis
Penetration depth in mm | 3 months after sinus augmentation
  measured through histomorphological analysis
Penetration depth in mm | 6 months after sinus augmentation
  measured through histomorphological analysis

CONTACTS AND LOCATIONS:
Overall Officials: Walther Wegscheider, Prof. DDr., Study Chair — Head of Department

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cordaro L, Bosshardt DD, Palattella P, Rao W, Serino G, Chiapasco M. Maxillary sinus grafting with Bio-Oss or Straumann Bone Ceramic: histomorphometric results from a randomized controlled multicenter clinical trial. Clin Oral Implants Res. 2008 Aug;19(8):796-803. doi: 10.1111/j.1600-0501.2008.01565.x. PMID 18705811
- [Background] Chiapasco M, Casentini P, Zaniboni M. Bone augmentation procedures in implant dentistry. Int J Oral Maxillofac Implants. 2009;24 Suppl:237-59. PMID 19885448
- [Background] Schopper C, Moser D, Sabbas A, Lagogiannis G, Spassova E, Konig F, Donath K, Ewers R. The fluorohydroxyapatite (FHA) FRIOS Algipore is a suitable biomaterial for the reconstruction of severely atrophic human maxillae. Clin Oral Implants Res. 2003 Dec;14(6):743-9. doi: 10.1046/j..2003.00959.x. PMID 15015951
- [Background] Ewers R. Maxilla sinus grafting with marine algae derived bone forming material: a clinical report of long-term results. J Oral Maxillofac Surg. 2005 Dec;63(12):1712-23. doi: 10.1016/j.joms.2005.08.020. PMID 16297691
- [Background] Scarano A, Degidi M, Perrotti V, Piattelli A, Iezzi G. Sinus augmentation with phycogene hydroxyapatite: histological and histomorphometrical results after 6 months in humans. A case series. Oral Maxillofac Surg. 2012 Mar;16(1):41-5. doi: 10.1007/s10006-011-0296-3. Epub 2011 Sep 24. PMID 21947545
- [Background] Kuhl S, Payer M, Kirmeier R, Wildburger A, Acham S, Jakse N. The influence of particulated autogenous bone on the early volume stability of maxillary sinus grafts with biphasic calcium phosphate: a randomized clinical trial. Clin Implant Dent Relat Res. 2015 Feb;17(1):173-8. doi: 10.1111/cid.12086. Epub 2013 May 28. PMID 23714235
- [Background] Raghoebar GM, Onclin P, Boven GC, Vissink A, Meijer HJA. Long-term effectiveness of maxillary sinus floor augmentation: A systematic review and meta-analysis. J Clin Periodontol. 2019 Jun;46 Suppl 21:307-318. doi: 10.1111/jcpe.13055. PMID 30624789